CLINICAL TRIAL: NCT00403728
Title: Protection by Ciclosporine A During Reperfused Acute Myocardial Infarction.
Brief Title: Ciclosporin A and Acute Myocardial Infarction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004.353
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Myocardial Infarction
Keywords: Ischemia; Reperfusion; Myocardial infarction; ciclosporin A; acute myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Ischemia

INTERVENTIONS:
Drug: ciclosporine A

SUMMARY:
Beyond its immunosuppressive properties, ciclosporine A (CsA) can also inhibit the opening of a mitochondrial mega-channel called the permeability transition pore (mPTP). Opening of the mPTP plays a key role in cardiomyocyte death during reperfusion following a prolonged ischemic insult. Ciclosporin A has been shown to reduce infarct size when administered at reperfusion in experimental models. The objective of the present study is to determine whether administration of CsA at reperfusion in patients with ongoing acute myocardial infarction treated by coronary angioplasty might reduce infarct size.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged more than 18, with suspected first acute myocardial infarction
* Within 12 hours of the onset of chest pain
* With a need for emergency revascularization by angioplasty. Patients must display a fully occluded (TIMI zero flow) culprit coronary artery, absence of visible collaterals and exhibit TIMI flow >2 after direct stenting by angioplasty.

Exclusion Criteria:

* Hypersensibility to ciclosporine A
* Cardiac arrest or cardiogenic shock
* Immunosuppressive disease (< 6 months): cancers, lymphomas, positive serology for HIV, hepatitis, etc.
* Known renal failure or serum creatinine > 120 µmole/l at admission
* Liver failure
* Uncontrolled hypertension
* Current pregnancy or women without contraception

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09

PRIMARY OUTCOMES:
Infarct size evaluated primarily by the area under the curve of CK and troponin I release over the first 72 hours of reperfusion.

SECONDARY OUTCOMES:
Myocardial contractile reserve assessed by dobutamine echocardiography at day 5.
No reflow evaluated by MRI at day 5
Recovery of myocardial contraction assessed by echocardiography and MRI at month 3

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ovize, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Michel Ovize, Lyon, France

REFERENCES:
- [Derived] Mewton N, Croisille P, Gahide G, Rioufol G, Bonnefoy E, Sanchez I, Cung TT, Sportouch C, Angoulvant D, Finet G, Andre-Fouet X, Derumeaux G, Piot C, Vernhet H, Revel D, Ovize M. Effect of cyclosporine on left ventricular remodeling after reperfused myocardial infarction. J Am Coll Cardiol. 2010 Mar 23;55(12):1200-1205. doi: 10.1016/j.jacc.2009.10.052. PMID 20298926